CLINICAL TRIAL: NCT02616107
Title: Improving Cancer Family Caregivers' Knowledge and Communication About Care Options
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Dena-Schulman-Green, Research Scientist, Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1407014318
Record Dates: First submitted 2015-11-18; First posted 2015-11-26 (Estimated); Last update posted 2017-03-07 (Actual); Status verified 2017-03

CONDITIONS: Family Caregivers
Keywords: Caregiver; Self-management; Care options; Goals of care; Breast cancer; Palliative care
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Family caregivers of breast cancer patients who consent to participate in the study have a 50/50 chance of being randomized to the intervention group and will receive the booklet, Managing Cancer Care: A Caregiver's Guide (MCC-CG) (N=18)
  Interventions: Other: Managing Cancer Care: A Caregiver's Guide
- Control (Active Comparator): Family caregivers of breast cancer patients who consent to participate in the study have a 50/50 chance of being randomized to the control group and will receive the Symptom Management Toolkit (N=17)
  Interventions: Other: Symptom Management Toolkit

INTERVENTIONS:
Other: Managing Cancer Care: A Caregiver's Guide — MCC-CG is a set of 7 printed modules including information about caregiver-nominated SM topics, conversation starters to facilitate communication with patients and providers, and links to caregiver resources. The modules are as follows:
  1. Becoming a Cancer Caregiver [role, changes, challenges, adjusting, self-care]
  2. Basics of Cancer Caregiving [physical, functional, emotional, social, & spiritual support; treatment timeline worksheet]
  3. Caregiver's Role in Managing Patient Care [who/what is involved; health care professionals worksheet]
  4. Managing Cancer Symptoms and Side Effects [common symptoms/side effects; maintaining health; nutrition & exercise; medication management worksheet]
  5. Care Options: [information on curative, palliative and hospice care]
  6. Talking About Goals of Care [information on goals of care conversations]
  7. Managing Transitions [defining transitions, transition examples, helping yourself and patient to manage transitions; transitions worksheet]
  Other Names: MCC-CG
  Arms: Intervention
Other: Symptom Management Toolkit — Along with an overview of symptom management, the Toolkit provides concise information on commonly experienced symptoms, including fatigue, alopecia, cognitive dysfunction, nausea and vomiting, and sleep problems, among others. Each chapter uses a question-and-answer format to cover the topics of who is most likely to experience the symptom, when and why the symptom may occur, how the symptom can be managed, and when to call a provider. Drs. Schulman-Green and McCorkle have previously tested the Symptom Toolkit in an attention-control group.
  Arms: Control

SUMMARY:
The purpose of this two-year mixed methods study is to develop and test an intervention to improve cancer family caregivers' knowledge of care options (curative, palliative, and hospice care) and goals of care communication as part of a self-management (SM) training program.

The two specific aims of this project are to:

1. Develop a psycho-educational intervention called Managing Cancer Care: A Caregiver's Guide (MCC-CG), for family caregivers of patients with breast cancer to increase knowledge of care options, goals of care communication, and other SM skills.
2. Evaluate the feasibility and preliminary efficacy of the MCC-CG in a pilot randomized controlled trial compared with an attention-control condition (symptom management education) on knowledge of care options, goals of care communication, and other key SM skills (engagement in SM, management of transitions and uncertainty, increasing self-efficacy, appropriate use of health care resources).

DETAILED DESCRIPTION:
The investigators will address and accomplish aim 1 by taking the following steps:

1. Conduct development focus groups with family caregivers of women with breast cancer.
2. Develop the MCC-CG intervention prototype.
3. Conduct feedback focus groups with family caregivers to evaluate the prototype.
4. Revise the MCC-CG.

To address and accomplish aim 2, the investigators will do the following:

1. Conduct a pilot RCT to evaluate the feasibility of recruiting and retaining a sample of family caregivers.
2. Assess the initial efficacy of the MCC-CG to improve knowledge of care options, goals of care communication, and other SM skills.
3. Estimate power and determine the best measures for a large RCT testing the MCC-PT and MCC-CG together.

ELIGIBILITY:
Inclusion Criteria:

* A family member of an individual with any stage of breast cancer receiving curative, palliative, or hospice care
* Aged 18+
* English speaking
* Live in Connecticut
* The patient for whom the participant is a caregiver has a six-month prognosis

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-07; Primary Completion 2016-11-09 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Knowledge of Care Options (KOCO) | 3 months
  11-item questionnaire in true/false format to assess knowledge of curative, palliative, and hospice care.
Medical Communication Competence Scale (MCCS) | 3 months
  Adjusted to reflect views of the family caregiver, the MCCS will assess participants' communication skills, including information seeking, providing, and verifying, and socio-emotional communication will be measured using the MCCS. Each item on the MCCS is presented with a Likert scale ranging from 7 (strongly agree) to 1 (strongly disagree).
Engagement in Cancer Self-Management Activities Scale (ECSMAS) | 3 months
  The 33-item ECSMAS was developed to measure cancer patients' self-reported self-management. The ECSMAS is organized around three conceptual domains derived from a metasynthesis of process of self-management in chronic illness: focus on illness needs, activating resources, and living with chronic illness. Items are adjusted to reflect views of the family caregiver, and an additional item has been added to the ECSMAS to assess caregivers' ability to manage transitions as a self-management skill (34 items total).

SECONDARY OUTCOMES:
Goals of Care Conversation | 3 months
  This form documents frequency, perceived quality, and content of goals of care conversations with patients and providers, as well as capturing any transitions experienced.
Caregiver Burden Scale (CBS) | 3 months
  This 22-item scale was developed to assess the experience of burden among caregivers, specifically addressing the dimensions of personal strain and role strain. Each item is presented with five response options ranging from 0-4 indicating "never", "rarely", "sometimes", "frequently", and "nearly always" sequentially.
Mishel Uncertainty in Illness Scale (MUIS) | 3 months
  Uncertainty will be measured using the 32-item MUIS, which was developed to measure the uncertainty adults perceive regarding symptoms, diagnosis, relationships, and planning for the future. Each item on the MUIS represents uncertainty in terms of a 5-point Likert-type format ranging from 1 (strongly disagree) to 5 (strongly agree). All items adjusted to reflect views of the caregiver.
Caregiver Competence Scale | 3 months
  Self-efficacy will be measured using a 4-point Likert scale, with four questions total.
Personal Gain Scale | 3 months
  Self-efficacy will be measured using a 4-point Likert scale, with four questions total.

OTHER OUTCOMES:
Demographic/Clinical form | Baseline
  Includes demographic data for caregivers and clinical data for the patient whom they provide care for.
Health Care Utilization | 3 months after 3-month data collection time point
  Data is abstracted from participants' medical records, including use of the emergency room, unscheduled hospital admissions, admission to ICU, use of chemotherapy and radiation in the last two weeks of life, and referral to hospice, among other indicators of disease burden as specified by the Center to Advance Palliative Care.

CONTACTS AND LOCATIONS:
Overall Officials: Dena J Schulman-Green, PhD, Principal Investigator — Yale School of Nursing
Locations (1):
- Smilow Cancer Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCorkle R, Ercolano E, Lazenby M, Schulman-Green D, Schilling LS, Lorig K, Wagner EH. Self-management: Enabling and empowering patients living with cancer as a chronic illness. CA Cancer J Clin. 2011 Jan-Feb;61(1):50-62. doi: 10.3322/caac.20093. Epub 2011 Jan 4. PMID 21205833
- [Background] Schulman-Green D, Ercolano E, Jeon S, Dixon J. Validation of the knowledge of care options instrument to measure knowledge of curative, palliative, and hospice care. J Palliat Med. 2012 Oct;15(10):1091-9. doi: 10.1089/jpm.2011.0514. Epub 2012 Jun 13. PMID 22694739
- [Background] Schulman-Green D, Jaser S, Martin F, Alonzo A, Grey M, McCorkle R, Redeker NS, Reynolds N, Whittemore R. Processes of self-management in chronic illness. J Nurs Scholarsh. 2012 Jun;44(2):136-44. doi: 10.1111/j.1547-5069.2012.01444.x. Epub 2012 May 2. PMID 22551013
- [Background] Grey M, Schulman-Green D, Knafl K, Reynolds NR. A revised Self- and Family Management Framework. Nurs Outlook. 2015 Mar-Apr;63(2):162-70. doi: 10.1016/j.outlook.2014.10.003. Epub 2014 Oct 15. PMID 25771190
- [Background] Schulman-Green D, Jeon S. Printed guide improves knowledge of curative, palliative, and hospice care among women with metastatic breast cancer. Support Care Cancer. 2013 Oct;21(10):2651-3. doi: 10.1007/s00520-013-1864-x. Epub 2013 Jun 1. No abstract available. PMID 23729228
- [Background] Schulman-Green D, Jeon S. Managing Cancer Care: a psycho-educational intervention to improve knowledge of care options and breast cancer self-management. Psychooncology. 2017 Feb;26(2):173-181. doi: 10.1002/pon.4013. Epub 2015 Nov 4. PMID 26537980
- [Background] Hinchey J, Goldberg J, Linsky S, Linsky R, Jeon S, Schulman-Green D. Knowledge of Cancer Stage among Women with Nonmetastatic Breast Cancer. J Palliat Med. 2016 Mar;19(3):314-7. doi: 10.1089/jpm.2015.0133. Epub 2016 Feb 8. PMID 26855201
- [Derived] Schulman-Green D, Linsky S, Blatt L, Jeuland J, Kapo J, Jeon S. Improving Breast Cancer Family Caregivers' Palliative Care Literacy: A Pilot Randomized Trial. J Fam Nurs. 2023 Feb;29(1):99-114. doi: 10.1177/10748407221099541. Epub 2022 Jun 7. PMID 35670155